CLINICAL TRIAL: NCT01983917
Title: Clinical Trial of Mobile Application to Enhance Diabetic Health Care
Brief Title: Mobile Application to Enhance Diabetic Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Irena Tsui, M.D., Assistant Professor of Ophthalmology, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-001117
Record Dates: First submitted 2013-10-30; First posted 2013-11-14 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; mobile application; diabetic retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Use of the Diabetes Application (Other)
  Interventions: Behavioral: Diabetes Mobile Application

INTERVENTIONS:
Behavioral: Diabetes Mobile Application

SUMMARY:
Prospective study to evaluate whether or not an internet application to coordinate and record diabetes management by the 1. diabetic patient/family caregiver 2. diabetic medical care team and 3. ophthalmology vision care team will decrease vision loss and blindness due to diabetic retinopathy. The aims will be measured through health psychology instruments to assess the effect of the application on management, motivation to control their disease, and commitment to comply with treatment. We will also measure objective health outcomes including Blood Pressure, Blood lipids level, hemoglobin A1c level, and Visual Acuity.

DETAILED DESCRIPTION:
This community-based study will involve the participation of healthcare professionals and physicians who are already treating the patient. Support and adequate training of the mobile application and the research protocol will be provided by the Study Coordinator.

The patient/family caregiver be asked to check their vision at home via their mobile application at regularly scheduled intervals as determined by their ophthalmologist. Patients will be expected to review postings of their visual acuity and office visits at a minimum of once a month intervals.

A staff member from the physician's office will post pertinent data from each office visit using a template. The ophthalmology template will include visual acuity, intraocular pressure, treatments given (if any), and uploaded retinal images. The non-ophthalmology physicians will post their office visit data in a free-form text box. Data entry can be performed by office staff and does not have to be done by a physician. Physicians will have access to view visual acuity records and physician postings from their own patients.

The research coordinator will collect health psychology data by administering validated health psychology questionnaires to assess patient depression, knowledge regarding diabetes and complications of diabetes, motivation to carry out diabetes care, reaction to increased knowledge of specific tests for diabetes and diabetic complications, and quality of life at 4-month intervals throughout the Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with diabetes mellitus and receiving care from either Jules Stein Eye Institute or the Gonda Diabetes Center at UCLA.
2. Between 14 and 75 years if age at the time of enrollment.
3. Internet access with Apple i-Phone, Apple i-Pad, and/or Apple i-Pod Touch on a weekly basis.
4. English language and Internet capability for data entry, monitoring, and comprehension of reports.
5. Able to attend Standard of Care visits for 1 to 3 years.
6. Able to understand and willing to sign the informed consent perform and comply with all study procedures

Exclusion Criteria:

1. Any social, mental or physical condition that impairs ability to give consent, maintain Internet access or attend physician visits.
2. Prior or concurrent eye or vision condition that would interfere with participation in or interpretation of the study.
3. Prior or concurrent disease or medical condition that is likely to compromise interpretation of the study.

3. Inability or unwillingness of the patient's diabetes medical care or ophthalmology vision care team to participate.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change of diabetic retinopathy risk factors | 1 year
  risk factors normalization by assessment of hemoglobin A1c percent, blood lipids level and blood pressure level as continuous variables.

SECONDARY OUTCOMES:
Motivation for adhering to treatment recommendations and follow-up | every 4 months
  Validated health psychology interments will be administer at enrollment and periodically during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Jules Stein Eye Institute, Los Angeles, California, United States